CLINICAL TRIAL: NCT05662735
Title: Randomized Controlled Trial of Laparoscopic Primary Diaphragm Repair With Sutures Alone Versus Sutures Reinforced With Mesh for Hiatus Hernia: A Long Term Follow-Up
Brief Title: Laparoscopic Primary Diaphragm Versus Mesh Repair for Hiatus Hernia: a Long-Term Follow-Up
Acronym: PRIME LTFU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Collaborators: Rijnstate Vriendenfonds (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL82840.100.22
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Hernia, Hiatal; Laparoscopic; Surgery; Recurrence; Mesh; Primary
MeSH Terms: conditions — Hernia, Hiatal; Recurrence

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant
Masking Description: Patients were blinded for repair with sutures alone or sutures with mesh augmentation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-absorbable sutures (Active Comparator): The hiatal hernia was corrected performing laparoscopic surgery. Primary repair of the hernia was done with non-absorbable sutures
  Interventions: Procedure: Suture repair
- Non-absorbable sutures and a TiMESH® (Active Comparator): The hiatal hernia was corrected performing laparoscopic surgery. Primary repair of the hernia was done with non-absorbable sutures and a TiMESH® to reinforce the repair.
  Interventions: Device: Mesh repair; Procedure: Suture repair

INTERVENTIONS:
Device: Mesh repair — Augmentation of hiatal hernia repair with TiMESH® reinforcement
  Arms: Non-absorbable sutures and a TiMESH®
Procedure: Suture repair — Primary laparoscopic repair of the hiatal hernia using non-absorbable sutures

SUMMARY:
Assessment of the recurrence of hiatal hernia five to ten years after repair using sutures versus sutures reinforced with non-absorbable mesh.

ELIGIBILITY:
Inclusion Criteria:

* Participant of the initial PRIME study
* Alive

Exclusion Criteria:

* No informed consent
* Additional hiatal hernia repair surgery during the follow-up period
* Pregnancy
* Patients that have stated they do not want to be approached for follow-up research

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of objective recurrence of a hiatal hernia | 5-10 years
  Objective measurement of the integrity of the hiatal hernia repair by CT-imaging

SECONDARY OUTCOMES:
Percentage of clinical recurrence of a hiatal hernia | 5-10 years
  Recurrence of symptoms related to a hiatal hernia measured by a questionnaire
Symptoms of gastroesophageal reflux disease | 5-10 years
  Percentage of participants that develop postoperative gastroesophageal reflux disease, measured by a questionnaire
Patient satisfaction | 5-10 years
  Overall satisfaction with surgical outcome measured by a questionnaire, on a scale from 0 to 10, where 0 means very unsatisfied with the outcome of the operation and 10 means very satisfied with the outcome of the operation. An additional question will be asked that assesses if the patient would undergo the operation again and can be answered by a simple 'yes' or 'no'.

IPD SHARING:
Plan to Share IPD: No